CLINICAL TRIAL: NCT05533749
Title: Improving Physical Health and Lifestyle Behaviors in Patients With Serious Mental Illness: a Cluster Randomized Controlled Trial on the Effectiveness of the Nurse-led GILL eHealth Intervention
Brief Title: Evaluating the Effectiveness of the GILL eHealth Intervention to Improve Physical Health and Lifestyle Behaviours in Patients With Severe Mental Illness
Acronym: GILL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Berno van Meijel, Prof. dr., Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL81729.029.22
Record Dates: First submitted 2022-08-25; First posted 2022-09-09 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Severe Mental Disorder; Metabolic Syndrome; Lifestyle; Somatic Screening; eHealth
MeSH Terms: conditions — Mental Disorders; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the intervention group or to care as usual. In the intervention group patients will receive the GILL eHealth intervention focusing on systematic somatic screening and lifestyle behaviours.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GILL eHealth module (Experimental): Patients will perform the GILL eHealth. This eHealth contains two modules focusing on systematic somatic screening and lifestyle behaviors.
  Interventions: Device: GILL eHealth
- Care as usual (No Intervention): Patients will receive usual care and have unrestricted access to mental care and treatment.

INTERVENTIONS:
Device: GILL eHealth — The aim of the successfully pilot-tested GILL eHealth intervention is to support mental health nurses and clinical nurse specialists in structured somatic screening and lifestyle promotion. The GILL eHealth intervention consists of two parts. Part one is OurGILL which focuses on systematic somatic screening and provides an overview of all somatic abnormalities. It promotes the prevention, early recognition and treatment of somatic problems. The second part is MyGILL. It provides the basis for drawing up a personalized lifestyle plan. The result of MyGILL is an overview of the performance of patients in different lifestyle areas. The eHealth intervention consists of an individual internet environment and is also supported by an app for mobile devices.
  Arms: GILL eHealth module

SUMMARY:
The aim of this study is to evaluate the effectiveness of the nurse-led GILL (Gezondheid in Lichaam en Leefstijl) eHealth intervention in patients with serious mental illness (SMI), compared to usual care. Expected is that the GILL eHealth intervention will be more effective than usual care in improving physical health and lifestyle behaviors. To evaluate this, we will perform a cluster randomized controlled trial with an embedded process evaluation of the implementation of the GILL intervention. 258 adult patients with serious mental illness and a body mass index of 27 or higher (overweight/obesity) will be included. The GILL eHealth intervention consists of two complementary modules for (a) somatic screening and (b) lifestyle promotion, resulting in a personalized somatic treatment and lifestyle plan. Trained mental health nurses and clinical nurse specialists will implement the intervention within the multidisciplinary treatment context, and will guide and support the patients in the promotion of their somatic health, including cardiometabolic risk management. The intervention will be compared to usual care, which includes treatment according to national guidelines. The outcome measures will be metabolic syndrome severity (primary), fitness, physical activity, lifestyle behaviors, quality of life, recovery, psychosocial functioning, health related self-efficacy and health care utilization after 1 year. The process evaluation focuses on the feasibility of the eHealth intervention, its acceptability for patients and health care providers (mainly mental health nurses and clinical nurse specialists), and barriers/facilitators to implementation.

ELIGIBILITY:
Inclusion Criteria:

* Meet the criteria of severe mental illness
* Aged from 18 to 65 years
* Body mass index (BMI) ≥ 27
* Access and ability to use internet
* Able and willing to sign informed consent

Exclusion Criteria:

* Contra-indications (to be assessed by the treating physician/psychiatrist) for participation due to acute psychiatric crisis or severe somatic diseases
* Subjects with a cognitive impairment sufficient to interfere with their ability to provide informed consent, complete study questionnaires, or participate in the intervention
* Pregnant or breastfeeding women at the time of inclusion
* Subject not able to communicate in the Dutch language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Metabolic Syndrome Severity Score (MSSS) | 12 months
  The MSSS includes the components sex, age, ethnicity, systolic blood pressure (mmHg), waistline circumference (cm), high-density lipoprotein, triglycerides and fasting blood glucose. A lower score is considered better.

SECONDARY OUTCOMES:
Weight (kg) | 12 months
  Weight is an indication for physical health.
Length (m) | 1 measurement
  Length will be measured to calculate the BMI.
Body Mass Index (kg/m2) | 12 months
  Body Mass Index (BMI) will be determined using the measured weight and length. A BMI between 18.5 and 25 is considered healthy.
Diastolic blood pressure (mmHg) | 12 months
  A healthy score of the diastolic blood pressure lies between 60 and 80 mmHg.
Lipid profiles (mmol/l) | 12 months
  LDL and total cholesterol will be determined. For the LDL a score below 3,0 mmol/l is considered good for healthy participants, participants with additional risks for cardiovascular diseases should have a score below 2.6 mmol/l, and for participants with a cardiovascular disease the score should be below 1.8 mmol/l. Overall, a lower LDL score is considered better. For the total cholesterol a score below 5.0 mmol/l is considered healthy.
HbA1c (mmol/l) | 12 months
  HbA1c is a measurement outcome to determine blood glucose. A score below 53 is considered healthy.
Six-minute walk test (6MWT) | 12 months
  The 6MWT is a measurement to assess physical fitness. It measures the walking distance in 6 minutes. A higher score indicates a longer distance walked and a better physical fitness.
International Physical Activity Questionnaire Short Form (IPAQ-SF) | 12 months
  The IPAQ-SF is a 10-item self-report questionnaire where participants recall the number of days and minutes of vigorous activity, moderate activity, walking and sitting time, over the past 7 days. A higher score indicates more physical activity.
Numeric Rating Scale (NRS) | 12 months
  The NRS will be used to determine the perceived physical health, physical activity and healthy eating of the past 4 weeks on a scale from 0-10. A higher score is considered better.
Short Form-12 | 12 months
  This is a generic, reliable and validated instrument to assess quality of life, containing 12 items derived from the Short Form 36 questionnaire. Physical and mental quality of life will be measured using the physical and mental component summary of the SF-12, respectively. A higher scores indicates a better health status.
Questionnaire about Processes of Recovery (QPR) | 12 months
  The QPR is a self-report 15-item questionnaire with a score range of 0-60 (QPR total). Higher scores are indicative of recovery.
Health of the Nation Outcome Scale (HoNOS) | 12 months
  The HoNOS is a clinician-rated instrument comprising twelve items on four domains (behavioral problems, organic problems, psychological symptoms, social problems), each item ranging from 0 (no problems) to 4 (severe problems). A lower score is considered better.
Patient Activation Measure (PAM-13) | 12 months
  The questionnaire assesses the participants' self-reported knowledge, skills and confidence for health-related self-efficacy. A higher score is considered better.

OTHER OUTCOMES:
Demographics | 12 months
  Age, gender, ethnicity, marital status, education level, employment status, psychiatric diagnoses, diagnosesof somatic diseases, current smoking status, number of years receiving mental care, and medication use.
Treatment Inventory of Costs in Patients with psychiatric disorders (TIC-P) | 12 months
  The TIC-P is a validated questionnaire designed for self-report in adult patients with a mental disorder to assess their utilization of the medical health care costs. The TIC-P items that will be used include 14 structured questions on the volume of medical costs, e.g. ambulatory services, private practice, and general practitioner. A higher outcome value means more health care costs.

CONTACTS AND LOCATIONS:
Locations (1):
- Parnassia Groep, The Hague, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will be intellectual property of the research team, and will be available for others in case of requests after publication of the results according to privacy regulations.

REFERENCES:
- [Derived] Hoogervorst MM, van Meijel B, Bruin EK, Beekman A, Boonstra N, Adriaanse M. The nurse-led GILL eHealth intervention for improving physical health and lifestyle behaviours in clients with severe mental illness: design of a cluster-randomised controlled trial. BMC Psychiatry. 2023 Sep 15;23(1):672. doi: 10.1186/s12888-023-05024-z. PMID 37715156